CLINICAL TRIAL: NCT03401697
Title: Curing HCV at Mount Sinai in Patients at High Risk for Disease Progression: HIV/HCV Co-infection and Type 2 Diabetes, New Solutions to the Challenge of Eliminating HCV
Brief Title: Eliminating Hepatitis C Virus
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Andrea Branch, Professor, Liver Diseases, Icahn School of Medicine at Mount Sinai
Other Study IDs: GCO 17-1070
Record Dates: First submitted 2018-01-09; First posted 2018-01-17 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Hepatitis C; HIV; Type2 Diabetes
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Blood (10 mL) will be collected from 100 HIV/HCV coinfected patients before and after HCV cure. sCD163 will be measured using the human CD163 Quantkine ELISA kit from R and D systems. Blood (10 mL) will also be collected from up to 50 patients who fail therapy or become reinfected with HCV. The HCV RNA quasispecies will be analyzed using the deep sequencing methods. Serum will be saved for HIV/HCV Co-infected.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HIV/HCV Co-infected: Patients with HIV/HCV co-infection
- Type 2 Diabetes: Patients with Type 2 Diabetes

SUMMARY:
Initially, HCV Informatics (C-IT) will be used to filter the EMR data of the one million people who receive care at Mount Sinai and identify candidates for HCV testing (baby boomers, patients with HIV infection) and candidates for HCV treatment (patients with positive test results for HCV RNA and no record of treatment).once treatment candidates have been identified through this proactive approach, their providers will be directly notified. HCV champions and patient navigators will be used to further lower barriers to the delivery of HCV care. They will be co-located at non-hepatology care sites and will help deliver open-label HCV treatment as part of standard medical care to 500 HIV/HCV co-infected patients and 200 patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for HCV treatment in patients with HIV/HCV co-infection

* 18 years of age or older
* HCV RNA positive
* Any HCV genotype
* Documented infection with HIV, with the following additional criteria: - Patients on HAART should be on a stable regimen for 4 weeks, with a CD4 count > 100, and an HIV viral load < 50 prior to initiation of HCV therapy Patients not on HAART should have a CD4 count > 350
* Expected life expectancy sufficient to receive a benefit from HCV cure
* No conditions that are contraindications for the use of HCV medications

Inclusion criteria for HCV treatment in patients with type 2 diabetes

* 18 years of age or older
* HCV RNA positive
* Any HCV genotype
* Documented diagnosis of type 2 diabetes, confirmed by medical record review by the study endocrinologist, Dr. Sherley Abraham
* Expected life expectancy sufficient to receive a benefit from HCV cure

Exclusion Criteria:

* No conditions that are contraindications for the use of HCV medications

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People who receive care at Mount Sinai and candidates for HCV testing or HCV treatment and co-located at non-hepatology care sites.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Change in the Number of Patients with sCD163 above the upper limit of normal | baseline and 3 years
  Change in the Number of Patients with sCD163 above the upper limit of normal at 3 years from baseline
Number of Type 2 Diabetes patients that initiate HCV treatment | 3 years
  The number of patients that initiate HCV treatment per month per patient navigator.

SECONDARY OUTCOMES:
sCD163 | 3 years
  blood sample for sC163, a marker of systemic inflammation.
Percentage of patients in need of repeated re-treatment | 3 years
  The percentage of patients in need of repeated re-treatment whose quasispecies analysis indicates that re-infection is the likely cause of recurrent HCV viremia. If such patients are identified, they will be referred for risk reduction counseling.
HOMA-IR | 3 years
  Homeostatic Model Assessment of Insulin Resistance (HOMA-IR). Healthy Range: 1.0 (0.5-1.4) Less than 1.0 means insulin-sensitive which is optimal. Above 1.9 indicates early insulin resistance. Above 2.9 indicates significant insulin resistance.
Number of resistance associated variant (RAV) | 3 years
  Resistance associated variant (RAV) testing from up to 50 patients who fail treatment or become re-infected
FIB-4 score | 3 years
  The FIB-4 score of HCV positive patients with type 2 diabetes. The Fibrosis 4 score is a non-invasive scoring system based on several laboratory tests that help to estimate the amount of scarring in the liver. This score has been studied in liver disease due to Hepatitis C and NASH. Formula : ( Age x AST ) / ( Platelets x ( sqr ( ALT )
HCV cure rate | 3 years
  The HCV cure rate among patients with type 2 diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Andrea D. Branch, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinia
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Direct outreach to providers (giving them the names of their patients who are candidates for treatment)